CLINICAL TRIAL: NCT04556123
Title: Bioimpedance Guided Management of Patients Scheduled for Transcatheter Aortic Valve Replacement: A Randomized Controlled Trial.
Brief Title: Management of Fluid Overload in TAVR
Acronym: EASE-TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Nitsche, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2074/2019
Record Dates: First submitted 2020-09-08; First posted 2020-09-21 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Volume Overload
Keywords: fluid overload; TAVR; decongestion; bioimpedance spectroscopy
MeSH Terms: conditions — Edema

STUDY DESIGN:
Intervention Model Description: Consecutive patients scheduled for TAVR fulfilling inclusion criteria will be enrolled. Patients with FO will be randomized in a 1:1 fashion to either BIS-guided decongestion or decongestion as per clinical judgement alone.
  Patients without FO will serve as an euvolemic control cohort.
Who Masked: Participant, Investigator
Masking Description: In order to avoid detection bias, FO patients in the non-BIS group as well as their treating physicians shall be blinded for BIS-results. Physicians and study participants will only be informed about the targeted dry body weight, if randomized to the BIS-guided decongestion group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fluid overload: BIS-guided decongestion (Experimental)
  Interventions: Other: Measurement of the hydration state and decongestive treatment according to bioimpedance spectroscopy
- Fluid overload: Decongestion based on clinical judgement (Active Comparator)
  Interventions: Other: Measurement of the hydration state and decongestive treatment according to clinical judgement alone
- No fluid overload: standard of care (No Intervention)

INTERVENTIONS:
Other: Measurement of the hydration state and decongestive treatment according to bioimpedance spectroscopy — The measurements will be performed in each center by a reference physician or nurse, using a portable whole body bioimpedance spectroscopy device, BCM (Fresenius Medical Care).
  The electrodes will be attached to one hand and one foot on the ipsilateral side, after the patient has been in the supine position for at least 5 minutes.
  Arms: Fluid overload: BIS-guided decongestion
Other: Measurement of the hydration state and decongestive treatment according to clinical judgement alone — Clinical judgement will be performed in each center by a reference physician or nurse
  Arms: Fluid overload: Decongestion based on clinical judgement

SUMMARY:
Fluid overload (FO) puts aortic stenosis (AS) patients at risk for heart failure and death. However, conventional FO assessment, including rapid weight gain, peripheral edema, or chest radiography, is inaccurate. Bioelectrical impedance spectroscopy (BIS) allows objective and reproducible FO quantification, particularly if clinically unapparent. FO as detected with BIS has recently been linked to worse clinical outcomes of AS patients undergoing transcatheter aortic valve replacement (TAVR).

It is the aim of the present randomised trial to evaluate the potential clinical benefit of pursuing an individualized decongestion treatment strategy in consecutive TAVR patients using BIS.

DETAILED DESCRIPTION:
This study is a randomized controlled trial investigating the effect of BIS-guided decongestive treatment on clinical outcomes in overhydrated patients scheduled for and receiving TAVR.

Centers participating in this trial are: Medical University of Vienna, Kepler University Hospital Linz

Consecutive adult patients with severe degenerative AS scheduled for TAVR will be prospectively enrolled at university-affiliated tertiary centers in Austria. Eligibility and decision for TAVR will be determined by a multidisciplinary Heart Team. All patients who are willing to participate will undergo assessment of volume status using BIS prior to intervention. Overhydrated subjects, defined as a relative fluid overload ≥7% (Rel. FO = fluid overload/extracellular water × 100%) and/or absolute fluid overload ≥1L as assessed by BIS, will then be randomly assigned to undergo BIS-guided pre- and postprocedural decongestion treatment vs. decongestion treatment based on mere clinical judgement of volume status in a 1:1 fashion. In order to avoid detection bias, FO patients in the non-BIS group as well as their treating physicians shall be blinded for BIS-results. Physicians and study participants will only be informed about the targeted dry body weight, if randomized to the BIS-guided decongestion group. Decongestion will be performed using standard medication (e.g. loop diuretics) and applied orally or intravenously, as appropriate. After TAVR, patients with FO will be followed before discharge from the hospital, after 3, 6 and 12 months.

Methods:

Patients will undergo standardized evaluation of their fluid status using a portable whole-body BIS device, the Body Composition Monitor (BCM, Fresenius Medical Care, Bad Homburg, Germany). Patients will be placed in supine position before the evaluation of their fluid status. Electrodes will be attached to the nondominant hand and the ipsilateral foot. Measurements will be conducted according to the manufacturer's manual. For each patient, only one bioelectrical impedance analysis will be performed, as this method has an adequate reproducibility. Fluid overload assessed by BCM is expressed as an absolute value in liters or as a relative value in %, calculated as the ratio between fluid overload (FO) and the content of extracellular water (ECW) and multiplied by 100 (Rel. FO = FO/ECW × 100%).

Prespecified study visits:

V0 (14+-13 days prior to TAVR): BIS measurement, pitting edema quantification, demographic factors, symptom assessment, cardiovascular risk factors, ECG, laboratory analysis (e.g. NT-pro BNP, hs-TnT), frailty assessment, KCCQ questionnaire, transthoracic echocardiography; V1 (90+-7 days post TAVR): BIS measurement, pitting edema quantification, demographic factors, symptom assessment, ECG, laboratory analysis (e.g. NT-pro BNP, hs-TnT), KCCQ questionnaire, transthoracic echocardiography; TV2 (telephone visit, 180+-7 days post TAVR): demographic factors, symptom assessment; V3 (360+-7 days post TAVR, =end of treatment): BIS measurement, pitting edema quantification, demographic factors, symptom assessment, ECG, laboratory analysis (e.g. NT-pro BNP, hs-TnT), KCCQ questionnaire, transthoracic echocardiography;

Outcome:

Cardiac outcomes (see below) will be assessed at 3 months (=prespecified interim analysis), and 12 months follwing TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years
* Scheduled TAVR for the treatment of severe aortic stenosis
* Fluid overlaod ≥7% and/or ≥1L by BIS prior to TAVR (necessary to undergo randomization process)

Exclusion Criteria:

* Unwillingness or inability to participate
* Pregnancy
* Chronic dialysis
* Severe electrolyte disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Hospitalization for heart failure and/or all-cause death | 3 and 12 months following TAVR

SECONDARY OUTCOMES:
Change from baseline to 12 months in KCCQ scores | 3 and 12 months following TAVR

OTHER OUTCOMES:
Change from baseline to 12 months in quantitative fluid levels | 3 and 12 months following TAVR
Change from baseline to 12 months in NT-proBNP levels | 3 and 12 months following TAVR
Change from baseline to 12 months in eGFR values | 3 and 12 months following TAVR

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nitsche, MD, Principal Investigator — Medical University of Vienna, Dpt. of Cardiology
Locations (2):
- Austria (2):
  - Karl Landsteiner University, Sankt Pölten, Lower Austria
  - Medical University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hong YA, Yoon HE, Choi BS, Shin SJ, Kim YS, Lee SY, Lee SH, Kim SH, Lee EY, Shin SK, Kwon YJ, Kim JH, Chang YK, Kim SY, Kim JE, Ahn SY, Ko GJ. The Effect of Strict Volume Control Assessed by Repeated Bioimpedance Spectroscopy on Cardiac Function in Peritoneal Dialysis Patients. Sci Rep. 2019 Nov 27;9(1):17679. doi: 10.1038/s41598-019-53792-0. PMID 31776362
- [Background] Machek P, Jirka T, Moissl U, Chamney P, Wabel P. Guided optimization of fluid status in haemodialysis patients. Nephrol Dial Transplant. 2010 Feb;25(2):538-44. doi: 10.1093/ndt/gfp487. Epub 2009 Sep 30. PMID 19793930
- [Background] Hur E, Usta M, Toz H, Asci G, Wabel P, Kahvecioglu S, Kayikcioglu M, Demirci MS, Ozkahya M, Duman S, Ok E. Effect of fluid management guided by bioimpedance spectroscopy on cardiovascular parameters in hemodialysis patients: a randomized controlled trial. Am J Kidney Dis. 2013 Jun;61(6):957-65. doi: 10.1053/j.ajkd.2012.12.017. Epub 2013 Feb 15. PMID 23415416
- [Background] Koell B, Zotter-Tufaro C, Duca F, Kammerlander AA, Aschauer S, Dalos D, Antlanger M, Hecking M, Saemann M, Mascherbauer J, Bonderman D. Fluid status and outcome in patients with heart failure and preserved ejection fraction. Int J Cardiol. 2017 Mar 1;230:476-481. doi: 10.1016/j.ijcard.2016.12.080. Epub 2016 Dec 21. PMID 28062131
- [Background] Stevenson LW, Perloff JK. The limited reliability of physical signs for estimating hemodynamics in chronic heart failure. JAMA. 1989 Feb 10;261(6):884-8. PMID 2913385
- [Background] Mulasi U, Kuchnia AJ, Cole AJ, Earthman CP. Bioimpedance at the bedside: current applications, limitations, and opportunities. Nutr Clin Pract. 2015 Apr;30(2):180-93. doi: 10.1177/0884533614568155. Epub 2015 Jan 22. PMID 25613832
- [Background] Nitsche C, Kammerlander AA, Koschutnik M, Sinnhuber L, Forutan N, Eidenberger A, Dona C, Schartmueller F, Dannenberg V, Winter MP, Siller-Matula J, Anvari-Pirsch A, Goliasch G, Hengstenberg C, Mascherbauer J. Fluid overload in patients undergoing TAVR: what we can learn from the nephrologists. ESC Heart Fail. 2021 Apr;8(2):1408-1416. doi: 10.1002/ehf2.13226. Epub 2021 Feb 13. PMID 33580746
- [Background] Nitsche C, Kammerlander AA, Koschutnik M, Dona C, Aschauer S, Sinnhuber L, Eidenberger A, Forutan N, Schartmueller F, Andreas M, Beitzke D, Bergler-Klein J, Bartko PE, Siller-Matula J, Winter MP, Anvari-Pirsch A, Goliasch G, Hengstenberg C, Mascherbauer J. Volume Status Impacts CMR-Extracellular Volume Measurements and Outcome in AS Undergoing TAVR. JACC Cardiovasc Imaging. 2021 Feb;14(2):516-518. doi: 10.1016/j.jcmg.2020.08.010. Epub 2020 Sep 30. No abstract available. PMID 33011120
- [Derived] Halavina K, Koschutnik M, Dona C, Autherith M, Petric F, Rockel A, Spinka G, Danesh D, Puchinger J, Wiesholzer M, Mascherbauer K, Heitzinger G, Dannenberg V, Koschatko S, Jantsch C, Winter MP, Goliasch G, Kammerlander AA, Bartko PE, Hengstenberg C, Mascherbauer J, Nitsche C. Management of Fluid Overload in Patients With Severe Aortic Stenosis (EASE-TAVR): A Randomized Controlled Trial. JACC Cardiovasc Interv. 2024 Sep 9;17(17):2054-2066. doi: 10.1016/j.jcin.2024.06.022. PMID 39260962